CLINICAL TRIAL: NCT06920407
Title: BreatheWell: Does Breathing Resistance Training Relax the Body and Calm the Mind?
Brief Title: BreatheWell: Train Your Breathing, Relax Your Body, Open Your Mind
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Paul Macey, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB #23-001177; 20233469 (Other Grant/Funding Number: Tiny Blue Dot Inc)
Record Dates: First submitted 2024-07-08; First posted 2025-04-09 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: Breathing; Stress; Breathing Training; Inspiratory Muscle Training; Breathing resistance training; Interoception; Physical and mental well-being; Health tracking; Oura
MeSH Terms: conditions — Respiratory Aspiration; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- IMT (Experimental): Participants will perform Inspiratory Muscle Training (IMT) using the PowerBreathe IMT K3 device at 65% resistance, focusing on the effects of higher resistance training on respiratory strength, physical well-being, and emotional well-being.
  Interventions: Device: Breathing training device (Inspiratory Muscle Training); Device: Oura Ring
- IMT Sham (Sham Comparator): Participants will perform the IMT procedure using the PowerBreathe IMT K3 device at 15% resistance to assess the effects of lower resistance on overall physical and emotional well-being, compared to higher resistance training.
  Interventions: Device: Breathing training device (Inspiratory Muscle Training); Device: Oura Ring
- Control (Active Comparator): Participants will not undergo the IMT procedure and will instead receive general health awareness through the Oura ring (a biometric ring and app), serving as the baseline group for comparison.
  Interventions: Device: Oura Ring

INTERVENTIONS:
Device: Breathing training device (Inspiratory Muscle Training) — Daily inspiratory muscle training (IMT) using the PowerBreathe IMT K3 device at varying resistance levels (15% for Sham and 65% for Experimental group) for 12 weeks. Participants will perform breathing exercises designed to assess the effects of different resistance levels on overall physical and emotional well-being, with a focus on how varying resistance impacts both respiratory strength and well-being.
  Other Names: Powerbreathe IMT K3 device
  Arms: IMT; IMT Sham
Device: Oura Ring — The Oura ring measures daily biometrics such as heart rate, sleep, and blood oxygen levels, providing personalized health data and insights. Participants have access to this data through a mobile app, allowing researchers to assess whether increased access to health data and awareness has an impact on overall physical and emotional well-being.
  Other Names: biometric ring

SUMMARY:
The goal of this study is to determine whether tasks related to breathing training (daily inspiratory muscle training (IMT) and increased access to health data/awareness) performed for 12 weeks leads to positive changes in mental and physical states, and if these changes are sustained three months later. The study will assess whether IMT, compared to a sham IMT and the control group, improves psychological well-being, body awareness, and physical relaxation. Although there is evidence that all three interventions make a difference, the extent of their impact is yet to be determined, so the study aims to compare the effectiveness of the interventions, aiming to determine which may be most beneficial.

The main questions the study aims to answer are:

* Do tasks related to breathing training (high resistance IMT, low resistance IMT, or access to health data) performed over 12 weeks enhance mental and physical well-being?
* Are the changes in mental and physical states sustained three months post-intervention?
* Is IMT more effective than sham IMT or simple health data engagement in improving well-being?
* Who benefits from each intervention?

Participants will be randomly assigned to three groups:

* IMT: Daily inspiratory muscle training at a moderate to high resistance.
* Sham IMT: Daily inspiratory muscle training at a low resistance.
* Control: Participants will track their health data but not engage in IMT.

Participants will:

* Engage in daily IMT or sham IMT training for 12 weeks.
* Engage with the Oura ring and app by checking in daily to sync the ring's data and review personal health insights.
* Complete daily and weekly surveys tracking mental and physical health.
* Have biometric data collected at baseline, post-intervention (12 weeks), and at a 3-month follow-up.

DETAILED DESCRIPTION:
This study seeks to investigate the impact of daily inspiratory muscle training (IMT) over 12 weeks on mental and physical well-being, focusing on whether the effects are sustained three months post-intervention. IMT is a breathing exercise known to improve respiratory function and reduce stress. This research will expand on previous findings showing that IMT can influence psychological states, such as increased awareness of the body, and improved relaxation and well-being. The investigators aim to compare the effects of IMT against a sham IMT group and a health data engagement-only group, assessing whether daily IMT enhances psychological well-being, body awareness, and physical relaxation.

Study Design and Groups:

* IMT Group: Participants will engage in daily inspiratory muscle training with the Powerbreathe device at moderate to high resistance, aimed at improving respiratory strength and exploring the effects of higher resistance training on well-being.
* Sham IMT Group: This group will complete daily IMT sessions at low resistance. This type of training encourages slower, deeper breaths, which some participants have found to help with relaxation and improving breath control.
* Engagement-Only Group: Participants will wear the Oura ring, which tracks health metrics such as heart rate, sleep, and physical activity. They will engage with the app to sync their data and review personal insights, fostering health awareness and self-monitoring.

Key Outcome Measures:

* Psychological Well-Being: Evaluated using the NIH Toolbox Psychological Well-Being (PWB) test.
* Body Awareness: Assessed with the Multidimensional Assessment of -Interoceptive Awareness (MAIA) scale.
* Physical Relaxation: Measured by heart rate variability (RMSSD), which reflects vagal tone and overall relaxation.

Study Procedures:

Participants will complete their assigned interventions for 12 weeks, with data collection at baseline, post-intervention (12 weeks), and at a 3-month follow-up. All participants will be asked to engage with weekly surveys to track their mental and physical health. The study also measures adherence, age, gender, physical activity, and sleep quality as potential confounding factors to better understand the broader impacts of the interventions.

This study aims to compare the effects of IMT at different resistance levels to see if it improves well-being, whether these benefits are maintained over time, and how it compares to simply engaging with health-tracking data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or higher
* Stable health for the past 3 months.

Exclusion Criteria:

* IMT contraindications which relate to people who should not raise lung, thoracic, or sinus pressures
* Current or recent (< 3 months) use of cardiovascular or psychotropic medications
* Diagnosed psychotic disorders
* Current participation in therapy
* Recent initiation of mind-body practice
* Current major illness or injury
* Regular use of personal tracking devices to monitor sleep, heart rate, activity, or related physiological data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Psychological Well-Being | From enrollment to the completion of the 12-week intervention period, followed by the observational period extending until week 24.
  Psychological well-being will be assessed using the NIH Toolbox Psychological Well-Being Scale. This instrument evaluates life satisfaction, positive emotions, and sense of purpose. Higher scores indicate greater psychological well-being.
  Unit of Measure: Standardized scale score
Change in Body Awareness | From enrollment to the end of the 12-week intervention period, followed by an observational period through week 24.
  Body awareness will be assessed using the Multidimensional Assessment of Interoceptive Awareness (MAIA), a validated questionnaire examining emotional awareness, body listening, and self-regulation. Higher scores indicate greater interoceptive awareness.
  Unit of Measure: Questionnaire scale score
Change in Heart Rate Variability (HRV) | From enrollment to the end of the 12-week intervention period, followed by an observational period through week 24.
  Heart rate variability will be assessed using the Root Mean Square of Successive Differences (RMSSD), reported in milliseconds. RMSSD reflects parasympathetic nervous system activity, with higher values indicating greater physiological relaxation.
  Unit of Measure: Milliseconds (ms)
Change in Inspiratory Muscle Strength | From enrollment (first physiology visit) to the end of the 12-week intervention period.
  Inspiratory muscle strength will be measured using the PowerBreathe training device and reported in centimeters of water pressure (cmH₂O), representing the pressure generated during inhalation against resistance.
  Unit of Measure: cmH₂O
Change in Peak Inspiratory Flow Rate | From enrollment (first physiology visit) to the end of the 12-week intervention period.
  Peak inspiratory flow rate will be measured using the PowerBreathe training device and recorded in liters per minute (L/min), indicating the maximum airflow achieved during inhalation.
  Unit of Measure: Liters per minute (L/min)
Change in Inhaled Volume per Breath | From enrollment (first physiology visit) to the end of the 12-week intervention period.
  Inhaled volume per breath will be assessed using the PowerBreathe training device and measured in milliliters (mL), indicating changes in lung capacity throughout the intervention.
  Unit of Measure: Milliliters (mL)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Macey, PhD, Principal Investigator — Professor
Locations (1):
- UCLA School of Nursing, Factor Bldg, 700 Tiverton Dr, Los Angeles, California, United States